CLINICAL TRIAL: NCT00901095
Title: Can Diet- & Exercise-induced Weight Loss Improve Asthma Control in Adults
Brief Title: Can Diet- and Exercise-Induced Weight Loss Improve Asthma Control in Adults?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Kaiser Permanente (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Associate Investigator, Palo Alto Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01HL094466 (NIH)
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual Care
- Lifestyle intervention (Experimental): The Lifestyle intervention group consists of in-person meetings co-led by an exercise specialist and dietician as well as follow-ups with an interventionist by phone.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Participants will attend a 15 weekly class sessions during the first 4 months. Classes will be co-lead by a dietician and exercise specialist and will involve a private weigh-in, a group discussion, a presentation of a lifestyle topic, 30 minutes of supervised moderate physical activity, followed by action-planning and goal-setting. During the next 2 months, participants will meet with a dietician on an individual basis for a private weigh-in, personal discussion and problem solving, review of self-monitoring records, and action-planning. The last 6 months will consist of applying and maintaining what has been learned in previous class sessions. Self-monitoring records, questions and problems will be discussed with interventions at least once every 2 months or more frequently if needed.
  Other Names: In-person sessions and self-monitoring
  Arms: Lifestyle intervention

SUMMARY:
The goal of the study is to investigate the efficacy of an evidence-based weight loss intervention, on a background of quality health care, on asthma control among obese adults. The intervention will employ a combination of recommended dietary and physical activity changes, and behavioral modification techniques.

ELIGIBILITY:
Inclusion Criteria:

Participants will meet all of the following:

* Age: 18-70 years of age;
* Obesity: BMI >30.0 kg/m2;
* Physician-diagnosed asthma that is poorly controlled:

  * Documented diagnosis of asthma on the current medical problem list
  * Currently prescribed an anti-asthma medication
  * Overall score <20 on the Asthma Control Test (ACT)64 or a score<3 on any of the first four ACT questions regarding symptoms, nighttime awakening, interference with normal activity, and SABA use for symptom relief
  * Demonstrable airway reversibility
* Seen in primary care at Kaiser at least once in the preceding 24 months;
* KPNC member for >1 year.

Exclusion Criteria:

Any of the following will exclude participants from the study:

* Inability to speak, read or understand English;
* Intermittent asthma, defined as either seasonal asthma or (daytime asthma symptoms < 2x/week and nocturnal symptoms < 2x/month and no use of long-term control medications);
* Diagnosis of COPD (emphysema or chronic bronchitis) on the current medical problem list or suggested by spirometry at baseline;
* Unwilling to attempt weight loss, including unwillingness to perform self-monitoring;
* Body weight change (+/-) > 10 pounds or use of weight-loss medications in the preceding 3 months;
* Inability to perform pulmonary function tests by spirometry in a consistent manner;
* Significant medical co-morbidities, including uncontrolled metabolic disorders (e.g., thyroid, diabetes, renal, liver), unstable heart disease, heart failure, and ongoing substance abuse;
* Diagnosis of psychiatric disorders that would limit adequate informed consent or ability to comply with study protocol;
* Regular use of medications that can cause weight gain (e.g., oral corticosteroids, insulin, certain oral hypoglycemics, certain antidepressants, etc.);
* Under treatment for cancer or another condition that may prevent completion of follow-up;
* Diagnosis of a terminal illness and/or in hospice care;
* Use of a pacemaker or other implanted medical devices;
* Pregnant, planning to become pregnant, or lactating;
* Actively enrolled in a care management program focused on weight loss at Kaiser or elsewhere;
* Already enrolled or planning to enroll in a research study that would limit full participation in the study or confound the observation and interpretation of the study's findings;
* Family household member already enrolled in the study;
* No longer receiving primary care from Kaiser, or planning not to do so within the study period;
* PCP determination that the study is inappropriate or unsafe for the patient;
* Investigator discretion for clinical safety or protocol adherence reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | Baseline, 6- and 12-months

SECONDARY OUTCOMES:
Lung function | Baseline, 6-, and 12-months
Quality of Life | Baseline, 6- and 12-months
Symptom-free days | Baseline, 6- and 12-month
Asthma-related and total health care utilization | Baseline, 6- and 12-month
BMI, diet, and physical activity | Baseline, 6- and 12-months
Adverse Events | 6- and 12-months
Patient Satisfaction | Baseline and 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D.,Ph.D., Principal Investigator — Palo Alto Medical Foundation
Locations (8):
- United States (8):
  - Kaiser Permananete, Fremont Medical Center, Fremont, California
  - Kaiser Permananete, Hayward Medical Center, Hayward, California
  - Kaiser Permananete, Novato Medical Center, Novato, California
  - Kaiser Permanente, Oakland, California
  - Kaiser Permanente, Richmond, California
  - Kaiser Permanente, San Francisco Medical Center, San Francisco, California
  - Kaiser Permananete, San Jose Medical Center, San Jose, California
  - Kaiser Permanente, Santa Clara, California

REFERENCES:
- [Derived] Xiao L, Lv N, Rosas LG, Au D, Ma J. Validation of clinic weights from electronic health records against standardized weight measurements in weight loss trials. Obesity (Silver Spring). 2017 Feb;25(2):363-369. doi: 10.1002/oby.21737. Epub 2017 Jan 6. PMID 28059466
- [Derived] Ma J, Strub P, Xiao L, Lavori PW, Camargo CA Jr, Wilson SR, Gardner CD, Buist AS, Haskell WL, Lv N. Behavioral weight loss and physical activity intervention in obese adults with asthma. A randomized trial. Ann Am Thorac Soc. 2015 Jan;12(1):1-11. doi: 10.1513/AnnalsATS.201406-271OC. PMID 25496399
- [Derived] Ma J, Strub P, Camargo CA Jr, Xiao L, Ayala E, Gardner CD, Buist AS, Haskell WL, Lavori PW, Wilson SR. The Breathe Easier through Weight Loss Lifestyle (BE WELL) Intervention: a randomized controlled trial. BMC Pulm Med. 2010 Mar 24;10:16. doi: 10.1186/1471-2466-10-16. PMID 20334686